CLINICAL TRIAL: NCT03036514
Title: Sublingual Sufentanil Tablet System (SSTS) Versus Intravenous Patient Controlled Analgesia (PCIA) With Morphine for Postoperative Pain After Back Surgery. A Single Center Case-control Study.
Brief Title: Sublingual Sufentanil Tablet System (SSTS) Versus Intravenous Patient Controlled Analgesia After Back Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Davina Wildemeersch, MD, University Hospital, Antwerp
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: 16/45/479
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Pain, Postoperative
Keywords: numeric rating scale; opioid side effects
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Single center case-control study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case (Experimental): Sublingual sufentanil tablet system (SSTS) for postoperative pain relief after laminectomy or spinal fusion in the first 72 hour period. Orange-coloured tablets containing 15mcg sufentanil, the patient-controlled device is designed to deliver a single tablet with a minimum lockout interval of 20 minutes.
  Interventions: Device: Sublingual sufentanil tablet system
- Control (Active Comparator): Patient-controlled intravenous analgesia (PCIA) for postoperative pain relief after laminectomy or spinal fusion in the first 72 hour period. This classic patient-controlled IV-pump contains 1mg/ml morphine and 50mcg/ml dehydrobenzperidol. Pump characteristics include 1ml each asked bolus, lockout interval of 8 minutes.
  Interventions: Drug: Patient-controlled intravenous analgesia

INTERVENTIONS:
Device: Sublingual sufentanil tablet system — Usage of a new patient-controlled SSTS in the postoperative phase after laminectomy or spinal fusion.
  Other Names: SSTS; Zalviso
  Arms: Case
Drug: Patient-controlled intravenous analgesia — Usage of classically used patient-controlled intravenous mophine-based postoperative analgesia after laminectomy or spinal fusion.
  Other Names: PCIA
  Arms: Control

SUMMARY:
In this study, numeric rating scale (NRS) and side effects are measured after usage of a sublingual sufentanil tablet system (SSTS) in comparison to intravenous patient controlled analgesia (PCIA).

DETAILED DESCRIPTION:
Sublingual sufentanil tablet system (SSTS) is compared in pain relief and side effect profile with the routinely used intravenous patient controlled analgesia (PCIA) with morphine in the postoperative phase after back surgery. The common use of PCIA with morphine is associated with a rather slow onset-time and active metabolites, with occurrence of potential harmful side effects as sedation and desaturation.

This mono-centric project involving American Society of Anesthesiologists (ASA) classification I-II patients undergoing elective neurosurgery (laminectomy) are recruited. Enrolled patients undergo numeric rating scale (NRS) and side effect questionnaire during the first 72h postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* scheduled elective laminectomy or spinal fusion
* American Society Anesthesiology Classification system (ASA) I-III

Exclusion Criteria:

* chronic opioid use (>3 months)
* pregnancy
* obstructive sleep apnea syndrome
* supplemental oxygen therapy at home
* postoperative use of non-steroidal anti-inflammatory or anti-neuropathic drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | 72 hours postoperatively
  Pain assessment by NRS

SECONDARY OUTCOMES:
Evaluation of side effect | 72 hours postoperatively
  Evaluation of pruritus, constipation, desaturation, nausea, vomiting, urine retention, hypotension, dizziness

CONTACTS AND LOCATIONS:
Overall Officials: Davina Wildemeersch, MD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- University hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No